CLINICAL TRIAL: NCT05296720
Title: EEG and Behavioral Correlates of Temporal Prediction in the Tactile Modality in Schizophrenia
Acronym: SchizPredicT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Psychothérapique de Nancy (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 021-A02434-37
Record Dates: First submitted 2022-02-17; First posted 2022-03-25 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2023-12

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients (Other): Patients with schizophrenia
  Interventions: Behavioral: Tactile stimulation
- Controls (Other): Controls matched with patients on age, sex and education level
  Interventions: Behavioral: Tactile stimulation

INTERVENTIONS:
Behavioral: Tactile stimulation — Participants are asked to react as fast as possible to a tactile stimulation

SUMMARY:
Patients with schizophrenia have disturbances in their sense of self, particularly their bodily self. Disorders of the sense of self are central to schizophrenia and are of interest because they are thought to be present prior to the development of the disorder, when only a few attenuated symptoms signal a risk of developing psychosis. Finding markers related to the sense of self would make it possible to predict which subjects, among those with minimal psychotic symptoms, will develop psychosis, and thus to better adapt management. Disturbances in the experience of the passage of time that accompany disturbances in the sense of self have been described particularly in subjects at risk of developing psychosis, and would predict the onset of the pathology. However, as with alterations in the sense of self, it can be difficult to get patients to describe their disturbances in the experience of time, and objective measures are required to facilitate detection of these disturbances. In the present protocol an objective measure of temporal perception mechanisms will be tested in relation to the sense of self.

The tests used in the protocol assess subjects' abilities to benefit from the passage of time and to use these abilities to predict and prepare for the occurrence of an event. The investigators have previously shown that patients with impaired bodily sense of self do not benefit from the passage of time to prepare themselves to process information in the future. The present protocol is aimed at developing a measure more sensitive to the patients' disorders by adding tactile measures.

DETAILED DESCRIPTION:
Patients with schizophrenia have disturbances in their sense of self, particularly their bodily self. Disorders of the sense of self are central to schizophrenia and are of interest because they are thought to be present prior to the development of the disorder, when only a few attenuated symptoms signal a risk of developing psychosis. Finding markers related to the sense of self would make it possible to predict which subjects, among those with minimal psychotic symptoms, will develop psychosis, and thus to better adapt management. Disturbances in the experience of the passage of time that accompany disturbances in the sense of self have been described particularly in subjects at risk of developing psychosis, and would predict the onset of the pathology. However, as with alterations in the sense of self, it can be difficult to get patients to describe their disturbances in the experience of time, and objective measures are required to facilitate detection of these disturbances. In the present protocol an objective measure of temporal perception mechanisms will be tested in relation to the sense of self.

The tests used in the protocol assess subjects' abilities to benefit from the passage of time and to use these abilities to predict and prepare for the occurrence of an event. The investigators have previously shown that patients with impaired bodily sense of self do not benefit from the passage of time to prepare themselves to process information in the future. The present protocol is aimed at developing a measure more sensitive to the patients' disorders by adding tactile measures.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female;
* Age between 18 and 60 years inclusive;
* Subject who has dated and signed the consent form (guardian or custodian prior to the commencement of any trial-related procedures if applicable);
* Enrolled in a social security plan or beneficiary of such a plan.

Exclusion Criteria:

* Psychoactive substance use disorders (as defined by DSM-V);
* Use of benzodiazepines (in the period prior to inclusion, for a duration equivalent to 5 half-lives of the product), cannabis (in the 2 months prior to inclusion; use of cannabis (THC) will be verified with a urine dipstick) or hallucinogenic substances (in the period prior to inclusion, for a duration equivalent to 5 half-lives of the product);
* Neurological pathology or sequelae;
* Attention deficit hyperactivity disorder (ADHD);
* A borderline personality disorder;
* Disabling sensory disorders;
* Person deprived of liberty or under court protection;
* Pregnant, parturient or nursing woman;
* Subject in a period of exclusion as defined by another clinical study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2023-04-13 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
measure of movement speed | month 2
  Motor anticipation: The participant moves his or her finger until a tactile stimulation is delivered, and the finger trajectory is recorded by means of a LED on the finger and a camera. The analysis of the trajectory allows for a measure of movement speed, acceleration and deceleration. The anticipation of the need to stop the movement is typically accompanied by a slowing down of the trajectory. The slowing down of the trajectory is used as a proxy for the anticipation of the tactile stimulation. We will measure at what time before the tactile stimulation the deceleration starts.

SECONDARY OUTCOMES:
Electroencephalographic measure | month 2
  The Electroencephalographic signal will be measured throughout the task in order to evaluate neurobiological correlates of the expectation. Expectation is associated with a CNV (Contingent Negative Variation), and this potential will be compared across the different experimental conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Anne GIERSCH, MD, PhD, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- Anne GIERSCH, Strasbourg, France